CLINICAL TRIAL: NCT02630121
Title: Effect of Oxymetazoline Hydrochloride in Combination With Fluticasone Propionate on the Apnea Hypopnea Index (AHI) in Subject With Persistent Nasal Congestion and Mild Obstructive Sleep Apnea. A Double Blinded Placebo Controlled, Crossover Prospective Trial.
Brief Title: Effect of Oxymetazoline Hydrochloride in Combination With Fluticasone Propionate on the Apnea Hypopnea Index (AHI) in Subject With Persistent Nasal Congestion and Mild Obstructive Sleep Apnea
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00001844
Record Dates: First submitted 2015-07-22; First posted 2015-12-15 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Sleep Apnea; Chronic Nasal Congestion
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Oxymetazoline; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo/Fluticasone Propionate (Placebo Comparator): Placebo Spray 2 Sprays QHS Fluticasone Propionate 1 spray BID
  Interventions: Drug: Placebo
- Oxymetazoline Hydrochloride /Fluticasone Propionate (Active Comparator): Oxymetazoline Hydrochloride 2 Sprays QHS Fluticasone Propionate 1 spray BID
  Interventions: Drug: Oxymetazoline Hydrochloride

INTERVENTIONS:
Drug: Oxymetazoline Hydrochloride — Proportion of the subjects with 50% reduction in AHI.
  Other Names: Afrin
  Arms: Oxymetazoline Hydrochloride /Fluticasone Propionate
Drug: Placebo — Proportion of the subjects with 50% reduction in AHI.
  Other Names: Nasal saline
  Arms: Placebo/Fluticasone Propionate

SUMMARY:
The addition of intranasal oxymetazoline for two weeks to already instituted optimal doses of intranasal fluticasone propionate will decrease the total number of obstructive apneas and hypopneas per hour of sleep in subjects with perennial allergic or non-allergic rhinitis and mild obstructive sleep apnea who have persistent nasal congestion despite maximum doses of NGCS.

DETAILED DESCRIPTION:
To evaluate the effectiveness of the addition of intranasal oxymetazoline to ongoing optimal doses of intranasal fluticasone propionate on the apnea/hypopnea index (AHI) in subjects with persistent nasal congestion and mild obstructive sleep apnea secondary to perennial allergic or non-allergic rhinitis despite treatment with the recommended doses of NGCS. The NOX T3 portable sleep monitor will be used to measure the AHI.

1. The Flow Sensor, as part of the NOX T3 portable monitor, will be used to assess flow limitation of the upper airway through calculation of the flattening index, a marker of upper airway resistance.
2. The Congestion Quantifier 7 (CQ7) questionnaire will be used to assess for an improvement in nasal congestion based on symptoms from the prior week.
3. The Nasal Congestion Visual Analog Scale (VAS) will be used to identify the changes in the severity of nasal congestion on a day to day basis.
4. The Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) will be used to assess the impact of perennial rhinitis and nasal congestion on activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 - 65 years of age.
2. At least a one year history of perennial allergic or non-allergic rhinitis.
3. Subjects must be on the maximum recommended doses of one of the following NGCS for at least one month. (See Table I)
4. AHI per hour of sleep > 5 and <15, minimum SpO2 88, indicating mild obstructive sleep apnea).
5. Average Nasal Congestion VAS of > 3-10 indicating moderate to severe nasal congestion between visits 1 and 2 based on daily symptoms (average of 7 scores).
6. Average Congestion Quantifier 7 score of 7 between visits 1 and 2 based on weekly symptoms (average of 2 scores).
7. Willingness to participate as indicated by signed informed consent.

Exclusion Criteria:

1. Presence of hypersensitivity to oxymetazoline or fluticasone propionate.
2. Subjects receiving allergen immunotherapy but not on a stable maintenance regimen for at least 30 days before the first study visit.
3. If the subject has perennial allergic rhinitis, he/she should not be entered into this study eight weeks before, during, or six weeks after any seasonal exacerbation.
4. Women who are pregnant or lactating.
5. Other known nasal diseases likely to affect deposition of oxymetazoline such as sinusitis, nasal polyps, or major nasal structural malformations.
6. Respiratory tract infections in the last 14 days.
7. Infections requiring antibiotics in the last 14 days.
8. Asthma or chronic obstructive pulmonary disease (COPD) requiring roflumilast or more than the recommended doses of inhaled corticosteroids, beta agonists, or antimuscarinic agents.
9. No systemic glucocorticosteroids for one month prior or during the study.
10. Cardiovascular disease with uncontrolled hypertension (BP160/80), arrhythmias and/or congestive heart failure.
11. Insulin-dependent diabetes mellitus and/or diabetic retinopathy.
12. Subjects with mild OSA (AHI 5-14) and SpO2 <88 for > 5 min during sleep that is identified during the screening portable sleep study.
13. Hypertension requiring more than two drugs, with the exception of hydrochlorothiazide, to achieve control.
14. A history of drug or alcohol abuse within the past 5 years.
15. Subjects who are currently abusing alcohol, illicit drugs, benzodiazepines, or narcotics.
16. Inability to cooperate, comply with study procedures or communicate with the investigator to successfully complete the study.
17. A history of benign prostate hypertrophy necessitating treatment.
18. A history of psychiatric problems which, in the opinion of the investigators, would impair participation in the study.
19. Subjects with a planned hospitalization during the study.
20. An infirmity, disability, or geographical location which seems likely to prevent regular attendance for subject visits.
21. Subjects with obstructive sleep apnea syndrome requiring CPAP therapy.
22. Subjects diagnosed with central sleep apnea (> 5 central events per hour) or moderate to severe OSA (AHI > 15) and SpO2 <88 for > 5 min during sleep identified during screening.
23. Use of the following medications within the time period specified below prior to Day -7 (Table 2).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects demonstrating a 50% reduction in the apnea hypopnea index after treatment with oxymetazoline hydrochloride and fluticasone propionate for 2 weeks. | 2 weeks
  This study is a double blinded, placebo control, cross over prospective trial. Each subject will complete the two arms in this study. The subject will be randomized to receive either oxymetazoline hydrochloride plus fluticasone propionate initially or placebo plus fluticasone propionate and complete treatment for a total of 2 weeks respectively. At the completion of each arm (prior to visit 3 and visit 5), the apnea hypopnea index will be measured.

SECONDARY OUTCOMES:
The proportion of subjects demonstrating an improvement in moderate to severe upper airway flow limitation as measured by a change in the flattening index after treatment with oxymetazoline hydrochloride and fluticasone propionate for 2 weeks. | 2 weeks
  This study is a double blinded, placebo control, cross over prospective trial. Each subject will complete the two arms in this study. The subject will be randomized to receive either oxymetazoline hydrochloride plus fluticasone propionate initially or placebo plus fluticasone propionate and complete treatment for a total of 2 weeks respectively. At the completion of each arm (prior to visit 3 and visit 5), upper airway flow limitation will be measured by a change in the flattening index from a value of ≥ 0.01 to 0.14 (moderate to severe airflow limitation) to a value of 0.15 - 0.3+ (mild airflow limitation to completely open upper airway).

OTHER OUTCOMES:
The proportion of subjects with a decrease in the severity of daily nasal congestion as measured by the Nasal Congestion VAS. | 7 weeks
  The proportion of subjects with a decrease in the severity of daily nasal congestion as measured by the Nasal Congestion VAS. Subjects will complete the Nasal Congestion VAS daily.
The Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) will be used to assess the impact of perennial rhinitis and nasal congestion on activities of daily living. | 6 weeks
  The Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) will be used to assess the impact of perennial rhinitis and nasal congestion on activities of daily living. Subjects will complete the questionnaire at visits 2, 3, 4, and 5 (total of 6 weeks).
The Congestion Quantifier 7 (CQ7) questionnaire will be used to assess for an improvement in nasal congestion based on symptoms. | 7 weeks
  The Congestion Quantifier 7 (CQ7) questionnaire will be used to assess for an improvement in nasal congestion based on symptoms from the prior week. Subjects will complete the questionnaire weekly for a total of 7 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Usf Asthma Allergy and Immunology Cru, Tampa, Florida, United States